CLINICAL TRIAL: NCT02997384
Title: Feasibility of Breast Cancer Risk Evaluation in Women From the General Population
Acronym: RIVIERA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A01082-49; 2016/2422 (Other: CSET number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Breastcancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- General practitioner
  Interventions: Other: Information
- gynecologist
  Interventions: Other: Information
- radiologist
  Interventions: Other: Information

INTERVENTIONS:
Other: Information — information of women about their risk of breast cancer and the screening methods recommended for them

SUMMARY:
This study aims to evaluate the feasibility (acceptability) of a consultation dedicated to informing women about their risk of breast cancer and the screening methods recommended for them according to the recommendations in force during a routine consultation at a general practitioner, a gynecologist or a radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Woman from 40 to 74 years old
* Understanding the French language

Exclusion Criteria:

Women will not be eligible for study if they are in any of the following situations:

* Cancer active or in the course of treatment type surgery, chemotherapy, or radiotherapy, whether breast or other organ
* Recent diagnosis <1 year of suspicious or cancerous lesions
* Psychiatric pathology not compatible with the study
* Poor understanding of the French language

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women 40 to 74 years seen in consultation by their attending physician, gynecologist or radiologist
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of women who agreed to measure their risk with personalized surveillance and screening recommendations during the consultation | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No